CLINICAL TRIAL: NCT05774600
Title: SSW Works: A Virtual Learning Environment for Occupational Skin Cancer Prevention Ph II
Brief Title: Virtual Sun Safe Workplaces Ph II (SSW Works)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0339; 4R44CA257778-02 (NIH)
Record Dates: First submitted 2023-02-09; First posted 2023-03-17 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Skin Cancer; Occupational Exposure
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSW Works (Experimental): SSW Works, is a virtual learning environment (VLE) for automated, comprehensive, on-demand, tailored distribution of the SSW program to private and public employers with outdoor workers. It will be delivered in both English and Spanish to managers and employees who work outdoors to reduce risk for skin cancer.
  Interventions: Behavioral: SSW Works
- Minimal Information Control (Active Comparator): Workplaces randomized to the control condition will receive a set of printed materials on occupational sun safety (1 mailing per year) as an attention control. These will include posters on personal protection and skin cancer incidence, risk assessment brochure, American Academy of Dermatology SPOT bookmark showing the ABCDEs of melanoma and skin self-examination, and a sun safety tip card from OSHA.
  Interventions: Behavioral: Minimal Information Control

INTERVENTIONS:
Behavioral: SSW Works — SSW Works is a behavioral, culturally tailored online intervention for skin cancer prevention amongst outdoor workers in the United States.
  Arms: SSW Works
Behavioral: Minimal Information Control — Provision of online materials for skin cancer prevention.
  Arms: Minimal Information Control

SUMMARY:
Americans who work outdoors are exposed to an extreme amount of solar ultraviolet radiation over a lifetime that substantially increases their risk for developing skin cancer. In Phase I, the feasibility of a virtual learning environment (VLE) for distributing the effective Sun Safe Workplaces (SSW) intervention to American employers will be established with input from senior managers and Hispanic and African American outdoor workers and development and evaluation of a prototype of the SSW Works VLE. In Phase II, the full SSW Works will be produced and tested for effectiveness at improving outdoor workers' sun protection in a randomized trial enrolling employers nationwide.

DETAILED DESCRIPTION:
Americans who work outdoors are exposed to an extreme amount of solar ultraviolet radiation (UV) over a lifetime that substantially increases their risk for developing skin cancer. Annually, skin cancer is diagnosed in over 3.5 million U.S. adults, melanoma kills nearly 7,000 Americans, and treatment costs at least $8 billion. The U.S. Surgeon General has identified occupational sun safety as a national priority. The team has spent the past two decades developing a successful comprehensive approach to occupational sun protection in 5 trials funded largely by the National Cancer Institute. Sun Safe Workplaces (SSW) combines policy and education to increase workplace actions on sun safety and employee sun protection practices. In this SBIR Fast-Track application, the investigators will develop a virtual learning environment (VLE), SSW Works, to distribute the SSW program to American workplaces. It will be comprised of a database, content management (interactive toolbox), and media platform (trackable training) that tailors the SSW program to management's readiness to innovate on sun safety based Diffusion of Innovations Theory. SSW Works will better integrate SSW into safety training by improving appropriateness for Hispanic and African American workers and conforming with the latest learning management systems technology (LMS). Strong scientific premise comes from the published literature and the team's 5 previous studies that demonstrated SSW is feasible and effective in public works, public safety, and outdoor recreation workplaces. The Phase I specific aims will establish the feasibility of SSW Works by 1) creating and validating an algorithm to tailor resources and implementation strategies to employers' stages in the diffusion of innovations process; 2) identifying unique attitudes, barriers, and practices related to sun safety among Hispanic and African American employees in focus group discussion and adjusting the SSW content; and 3) creating a prototype of the SSW Works VLE, including inputs, staging algorithm and tailored report, employee training compatible with a popular LMS, and storyboards of brief videos for managers and employees and testing it for feasibility and usability with managers and Hispanic and African American outdoor workers, and confirming that the training can operate within a popular LMS. In Phase II, SSW Works will be fully programmed and tested for effectiveness by achieving the specific aims of: 1) producing the full SSW Works, in English and Spanish, for distribution of the evidence-based SSW and 2) conducting a randomized controlled trial with 20 workplaces evaluating impact of SSW distributed over the SSW Works on employees' sun safety practices (primary outcome). The primary hypothesis is: compared to employers in the minimal information control group, employers assigned to receive SSW Works will have employees that practice more sun protection at posttest. The SBIR Fast-Track research is significant and innovative. SSW Works will have high impact and commercial potential because outdoor workforce is large and at very high risk for skin cancer, improving sun safety will reduce health care costs and save lives, and there are few commercial competitors.

ELIGIBILITY:
Inclusion Criteria:

* Manager Inclusion Criteria:
* Employed in a manager or supervisory position
* Responsible for worksite safety / health policy or education
* Read English or Spanish
* Consent to participate
* Complete the pre-test survey
* Employee Inclusion Criteria:
* Employed part-time / full-time at a participating employer
* Work at least 5 hours outdoors a week
* Read English or Spanish
* Consent to participate
* Complete the pre-test survey

Exclusion Criteria:

* Manager Exclusion Criteria:
* Read a language other than English or Spanish
* Employee Exclusion Criteria:
* Read a language other than English or Spanish
* Work exclusively indoors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Employee Sun Protection Practices at 1 year | Baseline assessment, 1 year assessment
  Employees will report frequency of sun protection at work (i.e., sunscreen with SPF 30+, long-sleeved shirts, long pants, hat with wide-brim, sunglasses, shade use, limit midday sun exposure, and have sunscreen, hat and eye protection at all times [1=never, 5=always]). SPF 30+ is advised in SSW to account for typical under-application that reduces effective SPF.
Change from Baseline Sunburn Prevalence at 1 year | Baseline assessment, 1 year assessment
  Employees will report prevalence of sunburn in past 3 months on the job (yes/no; number).

CONTACTS AND LOCATIONS:
Overall Officials: Mary Buller, MA, Principal Investigator — Kle
Locations (1):
- Klein Buendel, Golden, Colorado, United States